CLINICAL TRIAL: NCT01283269
Title: A Multicenter Rehabilitation Intervention for Amnestic Mild Cognitive Impairment
Brief Title: A Rehabilitation Intervention for Amnestic Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Mayo Clinic (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Melanie C Greenaway, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00034934; R01NR012419 (NIH)
Record Dates: First submitted 2011-01-11; First posted 2011-01-25 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Rehabilitation; Cognitive Intervention; Prevention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memory Support System or Computer (Experimental)
  Interventions: Behavioral: Memory Support System; Behavioral: Computer Training

INTERVENTIONS:
Behavioral: Memory Support System — Training in use of a memory notebook system
  Other Names: MSS
Behavioral: Computer Training — Computer brain fitness training
  Other Names: POSIT

SUMMARY:
Mild Cognitive Impairment (MCI) is often an early manifestation of Alzheimer's disease (AD). The ability to identify MCI has led to hope that health prevention models might work in AD as they have in cancer and heart disease. Interventions which help sustain functioning in MCI may delay progression to a clinical AD diagnosis. To date, interventions aimed at maintaining functioning in MCI have been pharmacologic in nature. The efficacy of these medications in MCI is controversial, and those with MCI are also often interested in other activities they can do to manage their memory loss.

When an individual is noted to have memory difficulties or MCI, a recommendation is often given for the patient to begin taking notes/using a calendar to help with memory or do cognitively stimulating activities. However, there is currently little instruction about how/what specific activities one should do and how effective they may be. The overall goal of this pilot project is to refine delivery of the Memory Support System (MSS)as a formal compensatory program for memory loss in MCI. Enrollment and retention data will be carefully investigated across 6 week and 10 day intervention groups. The investigators will compare participant adherence to the notebook training in the 6 week and 10 day versions of the intervention to the computer activity group. The investigators will also collect data on the clinical efficacy of the notebook and computer training to investigate if these interventions can sustain/improve functional level. Long term goals for this project also include delaying relocation for persons with MCI who may progress to dementia, thus not only improving the lives of these individuals, but also reducing health care expenditures.

The investigators will recruit a total of 60 individuals with MCI and their 60 program partners across all three sites for this project. At least 16 of these pairs will be recruited at Emory University (maximum of 20 pairs/40 individuals anticipated). The investigators will randomly assign participants to the 6 week notebook or computer training or 10 day notebook or computer training. All participants will also receive patient education regarding MCI and cognitive health.

Subsequent compliance with the MSS will be examined at 3 months, 6 months, and then annually following the intervention. Outcome measures will provide a detailed, multi-modal assessment of participants' functional level, overall cognitive functioning, mood, and self-efficacy, as well as caregiver burden and mood.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a research participant in the Alzheimer's Disease Research Center with a consensus diagnosis of amnestic Mild Cognitive Impairment (MCI: single domain or multi-domain).
* Has a program partner that has at least twice weekly contact with the participant
* Dementia Rating Scale-2nd Edition (DRS-2) score of 115 or greater
* Functional Ability Questionnaire (FAQ) score below 6.
* Program Partner with Mini Mental State Exam (MMSE) of 24 or greater. (If a program partner has an MMSE less than 24, the site PI will recommend that the person seek further evaluation of cognition through their primary care physician. The person with MCI will be encouraged to find an alternate program partner.)
* Either not taking or stable on nootropic(s) for at least 3 months
* Has English as primary language

Exclusion Criteria:

* Diagnosis other than amnestic MCI (single domain or multi-domain)
* Visual/hearing impairment or history of reading/writing disability sufficient to interfere with training
* Inclusion in another clinical trial that would exclude participation. Subject will be considered for participation at the end of such a trial or as appropriate.
* Baseline score on the self-report depression measure suggesting severe depression for either the participant or the program partner (>21 on the Centers for Epidemiological Studies - Depression Scale (CES-D) and need for psychiatric treatment. (If a patient or program partner has a CES-D greater than 21, the site Principal Investigator will rule out suicidal ideation and then recommend that the person seek further evaluation of mood from their primary care physician, psychiatrist, or other mental health practitioner. If they seek treatment and have been stable on that treatment for 3 months, they would then be allowed to be reconsidered for the study.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To assess participant adherence to Memory Support System (MSS) use at different levels (6 week, 10 day, or computer activity) of the training intervention. This will be measured by an overall adherence score (Adherence Assessment). | Baseline
To assess participant adherence to (Memory Support System) MSS use at different levels (6 week, 10 day, or computer activity) of the training intervention. This will be measured by an overall adherence score (Adherence Assessment). | Intervention End
To assess participant adherence to (Memory Support System)MSS use at different levels (6 week, 10 day, or computer activity) of the training intervention. This will be measured by an overall adherence score (Adherence Assessment). | 3 Month post intervention
To assess participant adherence to (Memory Support System) MSS use at different levels (6 week, 10 day, or computer activity) of the training intervention. This will be measured by an overall adherence score (Adherence Assessment). | 6 Months post intervention
To assess participant adherence to (Memory Support System) MSS use at different levels (6 week, 10 day, or computer activity) of the training intervention. This will be measured by an overall adherence score (Adherence Assessment). | 1 Year post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Greenaway, PhD, Principal Investigator — Emory University; Dona EC Locke, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Emory University, Atlanta, Georgia
  - Mayo Clinic-Rochester, Rochester, Minnesota